CLINICAL TRIAL: NCT06170580
Title: Improved Image Quality for Assessment of Carotid Artery Stenosis by Ultrafast Ultrasound FLOW Imaging
Acronym: CAS-iFLOW
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Collaborators: Netherlands Organisation for Scientific Research (Other Government)
Responsible Party: Sponsor
Other Study IDs: 114554
Record Dates: First submitted 2023-11-13; First posted 2023-12-14 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2024-11

CONDITIONS: Carotid Artery Stenosis
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Participants with a hemodynamic significant carotid artery stenosis
  Interventions: Diagnostic Test: Conventional duplex; Diagnostic Test: Ultrasound-based flow imaging using plane wave imaging; Diagnostic Test: Ultrasound-based flow imaging using cascaded wave imaging
- Participants without a hemodynamic significant carotid artery stenosis
  Interventions: Diagnostic Test: Conventional duplex; Diagnostic Test: Ultrasound-based flow imaging using plane wave imaging; Diagnostic Test: Ultrasound-based flow imaging using cascaded wave imaging

INTERVENTIONS:
Diagnostic Test: Conventional duplex — Conventional carotid duplex measurement
Diagnostic Test: Ultrasound-based flow imaging using plane wave imaging — Ultrasound-based flow imaging using plane wave imaging
Diagnostic Test: Ultrasound-based flow imaging using cascaded wave imaging — Ultrasound-based flow imaging using cascaded wave imaging

SUMMARY:
Objective: To evaluate the technical performance of a novel cascaded wave imaging technique compared to plane wave imaging for blood flow imaging in patients with and without carotid artery stenosis.

Study design: Observational, feasibility study in a total of 10 patients with and 10 patients without a hemodynamic significant carotid artery plaque.

Intervention (observational): all participants will undergo a carotid ultrasound measurement including conventional duplex ultrasound and ultrasound based flow imaging using plane waves and cascaded waves.

ELIGIBILITY:
Inclusion Criteria:

* Capacitated adult male or female (≥18 years old);
* Informed consent form understood and signed;
* Recent conventional duplex measurement of the carotid artery confirming either the absence or presence of a plaque

Exclusion Criteria:

* Hampered carotid blood flow imaging during conventional duplex/doppler measurements due to near to total carotid occlusion at the side of interest or a calcified plaque;
* History of radiation at the head-neck area;
* Participating in another clinical study, interfering on outcomes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 10 patients with and 10 patients without a hemodynamic significant carotid artery stenosis
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2023-11-16 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
2D velocity vector fields obtained by plane wave and cascaded wave imaging of the carotid artery | After study completion, average of one year

SECONDARY OUTCOMES:
Signal-to-noise ratio obtained from plane wave and cascaded wave imaging will be obtained and compared for different vessel depths | After study completion, average of one year
Cross-correlation maps of plane wave and cascaded wave imaging will be obtained and compared for different vessel depths | After study completion, average of one year
Velocity vector fields obtained from plane wave and cascaded wave imaging will be obtained and compared | After study completion, average of one year
Blood-flow related parameters, including vector complexity and vorticity, will be calculated from 2D velocity fields. | After study completion, average of one year
Spatiotemporal blood flow profiles obtained with plane wave, cascaded wave and conventional duplex ultrasound will be compared to assess the correlation between these techniques | After study completion, average of one year

CONTACTS AND LOCATIONS:
Locations (1):
- Radboud university medical center, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided